CLINICAL TRIAL: NCT05487846
Title: ADVANTAGE: Addressing Disparities for Veterans and African Americans Through Peer-Navigation for Testing and Genetic Evaluation
Brief Title: Peer Navigation for the Support of Metastatic Prostate Cancer Patients Undergoing Genetic Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21F.686; JT 17263 (Other: JeffTrial Number); PC200282 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Prostate Carcinoma; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Patient Navigation; Genetic Counseling; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (peer navigation) (Experimental): Patients receive assistance from a peer navigator during genetic evaluation processes. Peer navigators help patients schedule counseling appointments, discuss questions and concerns about testing, assist in sample collection, schedule a post-test disclosure visit, and do a results and recommendations debrief.
  Interventions: Behavioral: Patient Navigation; Other: Genetic Counseling; Other: Survey Administration
- Arm II (best practice) (Active Comparator): Patients receive standard care during genetic evaluation processes. Patients receive genetic counseling, undergo genetic testing, schedule a post-test disclosure visit, and receive their genetic test results and recommendations per standard care.
  Interventions: Other: Best Practice; Other: Genetic Counseling; Other: Survey Administration

INTERVENTIONS:
Behavioral: Patient Navigation — Receive peer navigation services
  Other Names: Patient Navigator Program
  Arms: Arm I (peer navigation)
Other: Genetic Counseling — Receive genetic counseling
  Arms: Arm I (peer navigation)
Other: Survey Administration — Ancillary studies
  Arms: Arm I (peer navigation)
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
  Arms: Arm II (best practice)
Other: Genetic Counseling — Receive genetic counseling
  Arms: Arm II (best practice)
Other: Survey Administration — Ancillary studies
  Arms: Arm II (best practice)

SUMMARY:
This clinical trial evaluates whether having a trained peer navigator helps African American men with prostate cancer that has spread to other parts of the body (metastatic) understand and navigate the genetic testing process better than not having a peer navigator. Genetic testing for men with prostate cancer is very important for making treatment and management decisions. However, understanding the risks, benefits, and steps of genetic counseling and testing can be very challenging for patients. African American men are especially less likely to participant in genetic testing due to lack of awareness or understanding, cultural beliefs, finances, or mistrust of the healthcare system. A peer navigator, someone who helps a patient through the information and the process, may be helpful to some men. This study evaluates whether having a peer navigator throughout the genetic evaluation process helps patients understand and engage in the process more.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop a peer-based navigation program for African American (AA) men with prostate cancer (PCA).

II. Conduct a pilot study of peer-navigated genetic evaluation vs. standard clinical care and assess feasibility of peer navigation.

SECONDARY OBJECTIVE:

I. Evaluating the intervention effects on decisional conflict and PCA genetics knowledge.

EXPLORATORY OBJECTIVE:

I. Assessing trust of the healthcare system and satisfaction with the genetic evaluation process.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive assistance from a peer navigator during genetic evaluation processes. Peer navigators help patients schedule counseling appointments, discuss questions and concerns about testing, assist in saliva collection, schedule a post-test disclosure visit, and do a results and recommendations debrief.

ARM II: Patients receive standard care during genetic evaluation processes. Patients receive genetic counseling, undergo genetic testing, schedule a post-test disclosure visit, and receive their genetic test results and recommendations per standard care.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* English speaking only
* Willing to comply with all study procedures and be available for the duration of the study
* Any individual >= 18 years old
* African American men who meet National Comprehensive Cancer Network (NCCN) criteria for testing will be offered participation. These criteria include any one of the following: (1) metastatic prostate cancer (PCA); (2) intraductal or ductal pathology; (3) T3a or higher; (4) grade group 4 or Gleason 8 or higher; (5) family history of breast, ovarian, prostate, pancreatic, colorectal, or uterine cancers in 3 or more blood relatives particularly if diagnosed at age < 50. These criteria have been adapted from the NCCN Prostate Cancer (version 2.2021) and NCCN Breast, Ovarian, and Pancreatic (version 2.2021) guideline

Exclusion Criteria:

* Patients that do not meet the inclusion criteria and children under the age of 18 will be excluded
* Anyone who has trouble understanding the consent or with significant anxiety detected during the consent process will also be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of pretest genetic counseling engagement | Up to 4 years
  Compared between randomized study groups. Tested using a chi-square test. Summarized between study groups in tables with descriptive statistics (e.g.'s, means and standard deviations if continuous, frequencies and percentages if discrete) with 95% confidence intervals and also graphically in data plots at each time they are assessed along with changes in responses over time.

SECONDARY OUTCOMES:
Mean changes in decisional conflict for genetic testing | Up to 4 years
  Compared between study groups over time. Summarized between study groups in tables with descriptive statistics (e.g.'s, means and standard deviations if continuous, frequencies and percentages if discrete) with 95% confidence intervals and also graphically in data plots at each time they are assessed along with changes in responses over time. Evaluated using mixed effects models with fixed effects for group indicator, time, and group-by-time interaction and random intercept effects for individual.
Mean changes in knowledge of cancer genetics | Up to 4 years
  Compared between study groups over time. Summarized between study groups in tables with descriptive statistics (e.g.'s, means and standard deviations if continuous, frequencies and percentages if discrete) with 95% confidence intervals and also graphically in data plots at each time they are assessed along with changes in responses over time. Evaluated using mixed effects models with fixed effects for group indicator, time, and group-by-time interaction and random intercept effects for individual.

OTHER OUTCOMES:
Healthcare system distrust | Up to 4 years
  Compared between two study arms. Summarized between study groups in tables with descriptive statistics (e.g.'s, means and standard deviations if continuous, frequencies and percentages if discrete) with 95% confidence intervals and also graphically in data plots at each time they are assessed along with changes in responses over time.
Satisfaction with the genetic evaluation process | Up to 4 years
  Compared between two study arms. Summarized between study groups in tables with descriptive statistics (e.g.'s, means and standard deviations if continuous, frequencies and percentages if discrete) with 95% confidence intervals and also graphically in data plots at each time they are assessed along with changes in responses over time.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Leader, DrPH, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No